CLINICAL TRIAL: NCT06565897
Title: Clinical Investigation to Assess the Efficacy of Manual Toothbrushes in the Reduction of Established Plaque and Gingivitis: a 6-week Clinical Study
Brief Title: Clinical Investigation to Assess the Efficacy of Manual Toothbrushes in the Reduction of Plaque and Gingivitis.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2024-04-MTB-FL-DR
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Plaque, Dental; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test regimen (Experimental): Brush with full ribbon toothpaste, 2x day / 2mins with paste & toothbrush provided
  Interventions: Drug: Test regimen
- Control regimen (Active Comparator): Brush with full ribbon toothpaste, 2x day / 2mins with paste & toothbrush provided
  Interventions: Drug: Control regimen

INTERVENTIONS:
Drug: Test regimen — toothpaste & manual toothbrush
  Arms: Test regimen
Drug: Control regimen — toothpaste & manual toothbrush
  Arms: Control regimen

SUMMARY:
Qualified subjects will be enrolled and randomized to one of the two study groups based on their initial Plaque and Gingivitis scores. Subjects will be instructed to use the products according to the instructions provided. Subjects will return to the dental office for evaluation after 1, 3, and 6, weeks of unsupervised product use at home. All subjects will be followed for adverse events throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects aged 18-70 years, inclusive.
* Availability for the six-week duration of the clinical research study.
* Good general health based on the opinion of the study investigator
* Minimum of 20 permanent natural teeth (excluding third molars).
* Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
* Initial mean plaque index of at least 0.6 as determined by Navy Plaque index.

Exclusion Criteria:

* Presence of orthodontic appliances.
* Presence of partial removable dentures.
* Tumor(s) of the soft or hard tissues of the oral cavity.
* Moderate and/or advanced periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study.
* Five or more carious lesions requiring immediate restorative treatment.
* Antibiotic use any time during the one-month period prior to entry into the study.
* Participation in any other clinical study or test panel within the one month prior to entry into the study.
* Dental prophylaxis during the past two weeks prior to baseline examinations.
* History of allergies to oral care/personal care consumer products or their ingredients.
* On any prescription medicines that might interfere with the study outcome.
* An existing medical condition that prohibits eating and/or drinking for periods up to 4 hours.
* History of alcohol and/or drug abuse.
* Self-reported pregnancy and/or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Plaque assessment | Initial reading, reading taken immediately following first brushing, 1-week, 3-weeks, and 6-weeks
  The dentition will be disclosed with disclosing solution and plaque scored according to the Refined Navy Plaque Index. Refinement of the Navy plaque index to increase plaque scoring efficiency in gum line and interproximal tooth areas.
Gingivitis Assessment | Initial reading, 1-week, 3-weeks, and 6-weeks
  A Loe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scoreable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror.

CONTACTS AND LOCATIONS:
Overall Officials: John Gallob, DMD, Principal Investigator — Consumer Research Consulting, LLC.
Locations (1):
- Consumer Research Consulting, LLC, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No